CLINICAL TRIAL: NCT00747227
Title: Clinical Evaluation of a Modified Light Transmission IOL
Brief Title: Safety and Efficacy of a Violet Visible Light Blocking Intraocular Lens (IOL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBLK-102-PRSM
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-10

CONDITIONS: Cataract
Keywords: cataract; monofocal; intraocular lens; acrylic
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZV9003 (Experimental): modified light transmission intraocular lens
  Interventions: Device: modified light transmission intraocular lens
- ZA9003 (Active Comparator): monofocal acrylic intraocular lens
  Interventions: Device: monofocal acrylic intraocular lens

INTERVENTIONS:
Device: modified light transmission intraocular lens — violet visible light blocking acrylic intraocular lens
  Other Names: ZV9003
  Arms: ZV9003
Device: monofocal acrylic intraocular lens — conventional hydrophobic acrylic intraocular lens
  Other Names: ZA9003
  Arms: ZA9003

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a new investigational modified light transmission monofocal intraocular lens compared to a conventional intraocular lens (IOL).

DETAILED DESCRIPTION:
The investigational IOL will be found to be safe and effective with respect to visual acuity, color vision, contrast sensitivity and complications and will be similar to results for the ZA9003 control eyes. Complication rates and adverse event rates will be within the FDA grid for posterior chamber IOLs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation has been planned
* Visual potential in both eyes of 20/30 Snellen or better after cataract removal and IOL implantation
* Preoperative corneal astigmatism of 1.5 diopters or less

Exclusion Criteria:

* Use of systemic or ocular medications that may affect vision
* Uncontrolled systemic or recurrent ocular disease
* Requiring an intraocular lens <15.0 or >26.0 diopters
* Abnormal results with the Farnsworth-Munsell D-15 and/or Ishihara color plates
* History of ocular trauma or prior ocular surgery
* Known pathology that may affect visual acuity or visual field
* Corneal abnormalities
* Pupil abnormalities
* Capsule or zonular abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger F. Steinert, M.D., Principal Investigator — University of California, Irvine, Dept. of Ophthalmology
Locations (11):
- United States (11):
  - Patrick Aiello, M.D., Scottsdale, Arizona
  - Randall E. Cole, M.D., Rogers, Arkansas
  - Aron Rose, M.D., New Haven, Connecticut
  - Y. Ralph Chu, M.D., Bloomington, Minnesota
  - Steven Silverstein, M.D., Kansas City, Missouri
  - Jon-Marc Weston, M.D., Roseburg, Oregon
  - William Christie, M.D., Cranberry Township, Pennsylvania
  - Mark Blecher, M.D., Philadelphia, Pennsylvania
  - Robert L. Bahr, M.D., Providence, Rhode Island
  - Vance Thompson, M.D., Sioux Falls, South Dakota
  - Jay Rudd, M.D., Lacey, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 250 subjects from normal cataract populations who were undergoing primary phacoemulsification with lens implantation and did not have any other visually significant ocular pathologies were selected at 12 investigation sites across the country
Groups:
- ZV9003 Intraocular Lens: modified light transmission intraocular lens
- ZA9003 Intraocular Lens: monofocal acrylic intraocular lens
Period: Overall Study
Arm/Group | ZV9003 Intraocular Lens | ZA9003 Intraocular Lens
Started | 126 | 124
Completed | 120 | 120
Not Completed | 6 | 4
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Illness | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZV9003 Intraocular Lens | ZA9003 Intraocular Lens | Total
Number analyzed (Participants) | 126 | 124 | 250
Age Continuous [Mean (Standard Deviation); unit: years] | 73.3 (8.0) | 71.5 (8.0) | 72.4 (8.0)
Age, Customized [Number; unit: participants]
  <60 years | 4 | 8 | 12
  Between 60 and 69 years | 35 | 41 | 76
  Between 70 and 79 years | 57 | 54 | 111
  >=80 | 30 | 21 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 68 | 146
  Male | 48 | 56 | 104
Region of Enrollment [Number; unit: participants]
  United States | 126 | 124 | 250

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Distance Visual Acuity
Description: Snellen Equivalent visual acuity of 20/40 or better
Time Frame: One year
Population: One subject was excluded from the analysis because the ZV9003 lens was implanted in the first eye and the ZA900 lens was implanted in the second eye. All subjects in the outcomes analysis had the same lens in both eyes.
Measure: Number; unit: participants
Arm/Group | ZV9003 Intraocular Lens | ZA9003 Intraocular Lens
Number analyzed (Participants) | 119 | 120
participants | 119 | 120

2. Secondary Outcome: Contrast Sensitivity
Description: Contrast sensitivity is the measurement of how faded an image may become before it can clearly be seen. Contrast sensitivity was measured in photopic and mesopic conditions at the following spatial frequencies: 3.0, 6.0, 12.0, and 18 cpd (cycles per degree). Contrast sensitivity is measured in log units. A higher value for the logarithmic units translates to better contrast sensitivity.
Time Frame: 4-6 months
Population: Binocular contrast sensitivity testing was reported for all binocular subjects with data available at the 4-6 month visit on 120 subjects in each group. One ZA9003 subject was tested at 3.0 cpd and not tested for 6.0 cpd through 18.0 cpd (mesopic and photopic). Testing for levels 6.0 through 18.0 were not reported.
Measure: Mean (90% Confidence Interval); unit: log contrast
Arm/Group | ZV9003 Intraocular Lens | ZA9003 Intraocular Lens
Number analyzed (Participants) | 120 | 120
log contrast
  Mesopic condition at 3.0 cpd | 1.62 [1.58 to 1.66] | 1.62 [1.58 to 1.66]
  Mesopic condition at 6.0 cpd | 1.65 [1.61 to 1.69] | 1.63 [1.58 to 1.68]
  Mesopic condition at 12.0 cpd | 1.14 [1.07 to 1.21] | 1.17 [1.10 to 1.24]
  Mesopic condition at 18.0 cpd | 0.60 [0.54 to 0.66] | 0.65 [0.59 to 0.71]
  Photopic condition at 3.0 cpd | 1.76 [1.73 to 1.79] | 1.74 [1.71 to 1.78]
  Photopic condition at 6.0 cpd | 1.91 [1.88 to 1.94] | 1.94 [1.91 to 1.98]
  Photopic condition at 12.0 cpd | 1.58 [1.54 to 1.62] | 1.59 [1.55 to 1.64]
  Photopic condition at 18.0 cpd | 1.09 [1.04 to 1.14] | 1.14 [1.09 to 1.19]

3. Primary Outcome: Uncorrected Distance Visual Acuity
Description: Snellen Equivalent of 20/40 or better at one year
Time Frame: One Year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | ZV9003 Intraocular Lens | ZA9003 Intraocular Lens
Number analyzed (Participants) | 119 | 120
participants | 110 | 116

4. Secondary Outcome: Subject Satisfaction - Subjects Satisfied With Overall Eyesight Rated as "Good" or "Excellent".
Description: Subjects indicating a subjective response to a multiple choice question, "At the present time, would you say your eyesight using both eyes (with glasses or contact lenses, if you wear them) is excellent, good, fair, poor, or very poor or are you completely blind?", on a multi-item questionnaire administered by interviewer to determine subject satisfaction with their overall visual outcome at the one year visit.
Time Frame: One Year
Population: Two subjects in the ZV9003 group did not complete the one year questionnaire.
Measure: Number; unit: participants
Arm/Group | ZV9003 Intraocular Lens | ZA9003 Intraocular Lens
Number analyzed (Participants) | 118 | 119
participants | 112 | 113

ADVERSE EVENTS:
Arm/Group | ZV9003 Intraocular Lens | ZA9003 Intraocular Lens
Serious Adverse Events (participants affected / at risk) | 1/126 | 1/124
Other Adverse Events (participants affected / at risk) | 0/126 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZV9003 Intraocular Lens (N=126) | ZA9003 Intraocular Lens (N=124)
Retinal Tear requiring secondary surgical intervention (Eye disorders) | 1 (1) | 1 (1) — Secondary surgical intervention required to repair adverse event of retinal tear. Principal Investigators felt it unlikely retinal tear was lens-related and both adverse events were reported as resolved with sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may not publish or disclose study data without Sponsor's prior written approval.